CLINICAL TRIAL: NCT05612087
Title: The Clinical Significance of Gut Permeability in Gastrointestinal Post Acute COVID-19
Brief Title: The Clinical Significance of Gut Permeability in Gastrointestinal Post Acute COVID-19 Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-09-010C
Record Dates: First submitted 2022-11-09; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Gastrointestinal Post Acute COVID-19 Syndrome
Keywords: post acute COVID-19 syndrome; gut permeability; Confocal laser endomicroscopy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — jejunum mucosa
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastrointestinal post acute COVID-19 syndrome: newly developped functional dyspepsia or irritable bowel syndrome after COVID-19 infection
  Interventions: Device: Confocal laser endomicroscopy

INTERVENTIONS:
Device: Confocal laser endomicroscopy — Confocal laser endomicroscopy at jejunum, duodenum and stomach

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) and the associated coronavirus disease 2019 (COVID-19) have been spreading all around the world for past 3 years. Some of these convalescent individuals experienced long- term sequelae termed 'long COVID', or 'post- acute COVID-19 syndrome'(PACS). Common manifestations are systemic, neuropsychiatric, cardio- respiratory and gastrointestinal [1].

The prevalence of gastrointestinal PACS was 2-5% in different literatures [2][3]. The risk factors of gastrointestinal PACS include anosmia, ageusia, and presence of chronic bowel disease, dyspeptic symptoms and the psychological comorbidity [4]. Previous articles have discussed pathogenesis of PACS, which was associated with increasing serum cytokine level and persisted inflammatory status [5]. Whereas, the influence of chronic inflammation to target organ has not been well studied. Liu et al explored the gut microbiota dynamics in patients with PACS, which revealed higher levels of Ruminococcus gnavus, Bacteroides vulgatus and lower levels of Faecalibacterium prausnitzii [6]. Another article established the association between multisystem inflammatory syndrome in children (MIS-C) and zonulin-dependent loss of gut mucosal barrier [7]. According to previous studies, infectious enteritis may cause subsequent post infectious irritable bowel syndrome [8][9], which was associated with increased gut permeability, T-lymphocyte, Mast cell and proinflammatory cytokine [10][11]. It is reasonable that gastrointestinal PACS might be also associated with dysfunction of gut mucosal barrier.

Confocal laser endomicroscopy (CLE) is a new endoscopic imaging tool that enables visualization of gut mucosa changes. The gut permeability could be accessed by CLE in patient with irritable bowel syndrome [12]. This study aimed to explore the association between gut permeability and gastrointestinal PACS.

ELIGIBILITY:
Inclusion Criteria:

* persisted gastrointestinal symptoms such as dyspepsia, abdomen pain, diarrhea or constipation 3 months after COVID-19 infection

Exclusion Criteria:

* Terminal cancer, surgical history of gastrointestinal tract, acute gastrointestinal tract bleeding, allergy to fluorescein, pregnant or breast feeding, helicobacter pylori infection, major cardiopulmonary disease, liver cirrhosis, end stage renal disease, autoimmune disease, inflammtory bowel disease, small intestinal bacterial overgrowth, celiac disease, type 1 diabetic mellitus, type II diabetic mellitus, gastroenteritis in 3 months, history of irritable bowel syndrome, usage of NSAID, steroid

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persisted gastrointestinal symptoms such as dyspepsia, abdomen pain, diarrhea or constipation 3 months after COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
gut permeability | 3 months
  leakage under Confocal laser endomicroscopy

SECONDARY OUTCOMES:
gut microbiome | 3 months
  fecal microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No